CLINICAL TRIAL: NCT01013168
Title: Clinical Study of OncoSorb® in Patients With Advanced Cancer Entities
Acronym: BP-005
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Achievement of feasibility and safety without achievement of clinical response.
Sponsor: BioPheresis GmbH (Industry)
Collaborators: Dr. M. Koehler GmbH (Unknown); ARTIMED Medical Consulting GmbH (Unknown)
Responsible Party: Niels Emmerich, Ph.D., CEO, BioPheresis GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-005
Record Dates: First submitted 2009-11-04; First posted 2009-11-13 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Advanced Cancer Entities
Keywords: OncoSorb; immune apheresis; sTNF-R1; sTNF-R2; sIL-2R; TNF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OncoSorb® column (Experimental)
  Interventions: Procedure: Apheresis using the OncoSorb column

INTERVENTIONS:
Procedure: Apheresis using the OncoSorb column — device is intended to specifically adsorb three soluble receptors (sTNF-R1, sTNF-R2 and sIL-2R α)
  Other Names: BioPheresis OncoSorb® system

SUMMARY:
The purpose of this study is to collect further data for safety and feasibility for the use of the medical device OncoSorb® in clinical routine for the treatment of patients with solid metastatic cancer entities who have failed standard therapies. OncoSorb® device is intended to specifically adsorb three soluble receptors (sTNF-R1, sTNF-R2 and sIL-2R α), which are known to inhibit the natural immune response of cancer patients mediated via tumor necrosis factor α (TNF- α).

DETAILED DESCRIPTION:
STUDY PURPOSE: The purpose of this study is to collect further data for safety and feasibility for the use of the medical device OncoSorb® in clinical routine for the treatment of patients with solid metastatic cancer entities who have failed standard therapies.

MEDICAL DEVICE: The medical device used in this clinical study is the OncoSorb® column. It is used with a specially modified Fresenius ART apheresis machine, associated tubing sets and an Albuflow plasma filter, also from Fresenius. These components comprise the extracorporeal immune apheresis system. The OncoSorb® column was CE certified in April 2008. The OncoSorb® device is intended to specifically adsorb three soluble receptors (sTNF-R1, sTNF-R2 and sIL-2R α), which are known to inhibit the natural immune response of cancer patients mediated via tumor necrosis factor α (TNF- α).

OBJECTIVES: Primary objective:

The primary objective is to evaluate the use of OncoSorb® therapy in clinical practice in terms of both safety and feasibility. This involves the evaluation of system-immanent issues (particularly occurrence of possible catheter infections and suitability of citrate/heparin anticoagulation) during the course of the clinical study prior the initiation of a phase II study.

Primary variables:

Occurrence of

* Possible catheter infection
* Suitability of citrate/heparin anticoagulation (with clogging of the extracorporeal circuit or bleeding as potential consequences)
* Adverse events/serious adverse events in general including changes of clinically relevant laboratory parameters, changes of vital signs, ECG changes)

Secondary objectives Evaluation of clinical efficacy as defined as objective response to treatment (according to RECIST), progression free survival (PFS), time to progression (TTP), clinical benefit, quality of life (QoL) and kinetics of soluble receptors.

Secondary variables:

* Objective response rate (ORR) to OncoSorb® therapy, defined as the proportion of patients with a confirmed CR or PR according to RECIST at efficacy evaluations I, II and III (after monthly Cycles 2, 4 and 6 and continuation until disease progression)
* Progression free survival (PFS)
* Time to progression (TTP)
* Clinical benefit of OncoSorb® therapy (defined as the proportion of patients with confirmed CR, PR and stable disease [SD]) in the evaluable patient population
* QoL (as assessed by EORTC QLQ-C30 rev. 3.0)
* Kinetics of sTNF-R1, sTNF-R2 and sIL-2R α (concentration levels pre-/post-apheresis as well as determination of receptor levels during treatments). Soluble receptor levels will be measured in the first 3 recruited patients at day 4 to 5 (hourly for the first 3 hours, every 2 hours for the following 6 hours and every 3 hours until treatment start on day 5).

STUDY POPULATION: A total of 5 evaluable patients will be recruited, aged 18 or older. Eligible patients will be identified at the NCT, Department of Medical Oncology or Department of Dermatology (Prof. Enk). Patient 5 will be a patient with cutaneous metastatic melanoma. One tumor lesion will be biopsied (tumor excision) in order to evaluate the induction of apoptosis triggered by TNF-α. The staging examination according to RECIST criteria will be conducted at the radiological department of the University of Heidelberg. Patients will receive a central venous catheter for the extracorporeal treatment at the site of Prof. Quentmeyer (St. Josefskrankenhaus, Heidelberg). The OncoSorb® treatment of the patients with OncoSorb® as extracorporeal immune apheresis device will be conducted either at the site of Prof. Rohmeiss (ze:ro dialysis center Schwetzingen) or at the site of Prof. Zeier (Nierenzentrum Heidelberg). For security reasons the recruitment of patients will be in consecutive order for patients 1 and 2: Patient 2 can be recruited only in the case that patient 1 has finalized OncoSorb treatments until the end of cycle 2. For the recruitment of subsequent patients (patients 3 to 5), no consecutive recruitment is planned. Patient 5 will optionally receive another biopsy (tumor excision) on day 5 of week 3 of the second treatment cycle to evaluate the biological effect of the OncoSorb treatment with respect to induction of apoptosis in response to TNF-α.

STUDY TREATMENTS: The study will start with a screening visit (day -21 to day 0) after obtaining informed consent of the patient. Patients screened for recruitment of patient 5 must give their consent for a baseline biopsy (tumor excision) and optional for a follow-up biopsy (after end of week 3 of cycle 2; tumor excision). Patients, who qualify for participation and are willing to participate, will receive in this period a central venous catheter for the conduction of the extracorporeal OncoSorb® therapy. During the treatment period all patients will receive OncoSorb® treatments consisting of daily immune adsorption treatment procedures 5 days per week for 3 weeks, followed by a resting period of one week. Due to safety reasons all patients will be hospitalized at the NCT during the first week of OncoSorb® treatment. Since currently no information exists about the counterregulation kinetics of sTNF-R1, sTNF-R2 and sIL-2Rα upon OnsoSorb® treatment, the collection of pharmacokinetic (PK) data is planned for the first 3 recruited patients. Blood samples for PK measurements of these patients will be taken between day 4 and 5 of the first treatment cycle under hospitalized conditions. PK data will be essential for designing an optimized treatment schedule (potential reduction of both frequency and apheresis time) of subsequent patients on trial. The schedule of the first 3 patients constitutes a one monthly treatment cycle. For the 2 remaining patients of this study the treatment plan will be re-designed according to the PK data obtained from the first 3 patients on treatment. The efficacy evaluation will be carried out 8 weeks after beginning of treatment. Patients with progression of disease may be withdrawn from OncoSorb® treatment. Patients with complete response (CR), partial response (PR) or stable disease (SD) will be offered to continue OncoSorb® treatments until disease progression. In this case efficacy evaluation (CT scans) will be performed every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic solid cancer who have documented progressive disease and who have failed standard therapy
* Measurable disease (RECIST criteria)
* Expected survival of at least 4 months
* Performance status ECOG 0 and 1
* Vital laboratory parameters within normal range, or protocol specified ranges
* Able to give written informed consent
* The patient's sTNF-R1, sTNF-R2 levels in citrate plasma are > 500 pg/ml and > 1000 pg/ml respectively
* The patient has adequate renal function as evidenced by glomerular filtration rate > 80 ml/min
* Patient 5 with metastatic melanoma must have skin lesion(s)
* Patient 5 with metastatic melanoma should have slow tumor progression
* Patient 5 with metastatic melanoma must have an intact TNF-receptor signaling cascade, resulting in measurable induction of cancer cell apoptosis following the exposition to TNF-α in vitro. This will be evidenced by destruction of primary autologous cancer cells obtained by biopsy.

Exclusion Criteria:

* Other serious or significant illnesses
* Other malignancy within the last 3 years, except for target oncological indication (does not exclude metastatic sites)
* Known immunodeficiency
* Known HIV or hepatitis positivity
* Using systemic immunosuppressive drugs. (Exceptions: Specific COX-2 inhibitors; low dose aspirin for cardiovascular event prevention; topical/inhaled steroids)
* Chemotherapy, immunotherapy or radiotherapy within two weeks prior to start of OncoSorb® treatments provided that all prior therapy related toxicities are resolved
* Participation in a prior clinical trial involving an investigational agent within the last 2 weeks
* Not available for clinical follow-up assessments
* Pregnancy or breastfeeding
* Refusal or inability to use effective means of contraception for women of childbearing potential
* Mental impairment that may compromise ability to give informed consent and to comply with study requirements
* History of a myocardial infarction within 6 months prior to the start of study, uncontrolled congestive heart failure, or any current Grade 3 or 4 cardiovascular disorder despite treatment
* Coagulation disorders and / or a history of thromboembolic complications
* Any significant disease that, in the Investigator's opinion, should exclude the patient from the study
* Known hypersensitivity or allergy to rabbit proteins
* Known hypersensitivity to heparin or citrate
* The patient receives Angiotensin-Converting Enzyme (ACE) inhibitors or Coumadin (Marcumar®) as concomitant medication
* Patient 5 with metastatic melanoma with brain metastases (MRT scan)
* Patient 5 with metastatic melanoma is severely immunocompromised (patient must have average or low TREG counts, no dysfunctional T cells like e.g. CD28-)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of: possible catheter infection, suitability of citrate/heparin anticoagulation, adverse events/serious adverse events in general | 0-6 months

SECONDARY OUTCOMES:
Overall response defined by RECIST criteria | 8 week response rate
Quality of life questionaire (as assessed by EORTC QLQ-C30 rev. 3.0) | 0-6 months
Kinetics of sTNF-R1, sTNF-R2 and sIL-2R α | receptor levels will be measured on treatment day 4

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Krauss, MD, Principal Investigator — Nationales Centrum für Tumorerkrankungen (NCT); Niels Emmerich, PhD, Study Director — BioPheresis GmbH
Locations (6):
- Germany (6):
  - St. Josefskrankenhaus, Heidelberg, Baden-Wurttemberg
  - Dermatologische Onkologie am NCT, Heidelberg, Baden-Wurttemberg
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg, Baden-Wurttemberg
  - Nierenzentrum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinik Heidelberg - Diagnostische und Interventionelle Radiologie, Heidelberg, Baden-Wurttemberg
  - ze:ro Dialysezentrum Schwetzingen, Schwetzingen, Baden-Wurttemberg

REFERENCES:
- See also: BioPheresis OncoSorb® product homepage — http://www.biopheresis.de/index.php?id=8